CLINICAL TRIAL: NCT04421573
Title: Cervical Plexus Hydrodissection With D5W for PTSD Versus Delayed Treatment/Usual Care
Brief Title: Cervical Plexus Hydrodissection With D5W for PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Dean Reeves Clinic (Other)
Collaborators: Paul Johnson, D.O. (Unknown); Eric Phillippi, M.D. (Unknown); Ryan Wood, N.D. (Unknown); Danesh Mazloomdoost (Unknown)
Responsible Party: Principal Investigator, Dr. Dean Reeves, Principal Investigator, Dr. Dean Reeves Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DextrosePTSD1
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: PTSD
Keywords: Dextrose; Hydrodissection; Cervical Plexus
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Randomized open-label crossover study comparing BHDCP with D5W versus a waiting period in which usual care is allowed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCPHD-D5W with usual care (Experimental): Bilateral cervical plexus hydrodissection with D5W (BCPHD-D5W) at 0, 2, 4, and 8 weeks.
  All helpful treatment methods already underway are continued. Other new treatment methods are discouraged.
  Interventions: Procedure: BCPHD with D5W
- Waiting period with usual care (Active Comparator): All helpful treatment methods already underway are continued. Other new treatment methods are discouraged.
  Interventions: Procedure: Waiting period with usual care

INTERVENTIONS:
Procedure: BCPHD with D5W — D5W is injected under the investing fascia of the sternocleidomastoid muscle (SCM) using ultrasound guidance in order to infiltrate the space containing the cervical plexus. This is performed on both sides.
  Arms: BCPHD-D5W with usual care
Procedure: Waiting period with usual care — Same as previous group description
  Arms: Waiting period with usual care

SUMMARY:
PTSD is a chronic mental health condition that drastically reduces an individual's quality of life Dextrose injection with a small needle has been used for chronic pain patients and observational results have shown it to be effective in reducing anxiety, brain fog, and depression in patients with PTSD. This randomized trial will compare dextrose injection with a delayed/usual treatment control.

DETAILED DESCRIPTION:
PTSD is a well-recognized debilitating mental health condition associated with previous trauma exposure. It is part of the DSM-5 Trauma and Stressor related disorders category. Treatments for PTSD normally involve a multi-disciplinary approach. First-line treatments include psychotherapy and serotonergic reuptake inhibitors. Many patients fail pharmacotherapy and psychotherapy. Unilateral stellate ganglion block performed favorably for treatment of PTSD in a recent RCT, based upon an expectation that the cervical sympathetic system is neuropathically upregulated in PTSD. However, inclusion of lidocaine requires the presence of an emergency response team due to the potential for inadvertent intravascular injection with generalized seizures or hypotension, and inadvertent laryngeal or phrenic nerve block. Perineural injection of peripheral nerves, plexi, or sympathetic ganglia with dextrose 5% in water (D5W), has performed well empirically in the treatment of post-traumatic stress disorder. No lidocaine is utilized, which allows for avoidance of lidocaine toxicity risk, or any risk of nerve block. Because of that, bilateral procedures are feasible, and these procedures can be performed in any outpatient office with ultrasound availability, as emergency team backup is not necessary, making the procedure readily accessible. A cumulative benefit has been observed, as well. The effects of BHDCP with D5W as a stand-alone treatment for PTSD has not been formally evaluated. This small study is designed as a feasibility study with study acceptance rate, protocol adherence, and satisfaction as primary outcomes. Secondary outcomes will include short term and long-term effects of BHDCP with D5W on the Post Traumatic Stress Disorder Check List for Civilians (PCL-C), The primary hypotheses are that the acceptance rate and protocol adherence will both exceed 80%, and satisfaction will be 6/10 or higher on a 0-10 satisfaction scale. A study size of 24 is planned, based on power analysis.

ELIGIBILITY:
Inclusion Criteria:

* Not involved in another study of PTSD treatment
* Reliable transportation
* Comfortable with computers
* Tried 2 or more medications for treatment of PTSD symptoms
* Tried 2 or more non-medication treatments for PTSD symptom
* No known life-threatening illness
* Not taking daily narcotics
* Not having 3or more alcoholic drinks on an average day
* No active suicidal plans
* No major surgery plans
* No major life stress that might interfere with completing study
* Symptoms for more than 1 year
* Not planning to move for next 18 months.
* Living within an hour of Portlland, OR, Madison, WI, or Lexington, KY
* Wiling to provide 2 email and 2 phone contact methods
* Willing to answer questions on multiple occasions over the course of a year.
* Willing to be assigned to 3 months of usual care treatment
* No diagnosis of schizophrenia, Borderline Personality Disorder, or Bipolar Disorder.
* No severe needle phobia
* Chronic pain ≤ 5/10
* PCL-C score ≥ 50

Exclusion Criteria: None separate from inclusion criteria

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Consent rate | 3 months
  Percentage consent rate for qualifying participants
Data Capture rate | 3 months
  Percentage data capture
Satisfaction rating | 3 months
  Satisfaction with treatment outcome as measured by a 0-10 Numerical Rating Scale (NRS)

SECONDARY OUTCOMES:
PCL-C Score | 3 months
  Improvement (reduction) in PTSD check list for civilians
HADS scale | 3 months
  Improvement in the Hospital Anxiety and Depression Scale
EuroQOL 0-100 | 3 months
  0-100 rating of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D Reeves, M.D., Principal Investigator — Dr. Dean Reeves Clinic
Locations (4):
- United States (4):
  - Danesh Mazloomdoost, Lexington, Kentucky
  - Paul W. Johnson, D.O., Clinic., Portland, Oregon
  - NW Regen, Tigard, Oregon
  - Eric Phillippi M.D. Clinic, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rae Olmsted KL, Bartoszek M, Mulvaney S, McLean B, Turabi A, Young R, Kim E, Vandermaas-Peeler R, Morgan JK, Constantinescu O, Kane S, Nguyen C, Hirsch S, Munoz B, Wallace D, Croxford J, Lynch JH, White R, Walters BB. Effect of Stellate Ganglion Block Treatment on Posttraumatic Stress Disorder Symptoms: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Feb 1;77(2):130-138. doi: 10.1001/jamapsychiatry.2019.3474. PMID 31693083